CLINICAL TRIAL: NCT02701686
Title: A Comparison of the Effectiveness of Two Approaches (Quit Immediately: QI and Cut Down to Quit: CDTQ) in Achieving Smoking Abstinence Among Patients Having Follow-up in a GOPC: A Pilot Randomized Controlled Trial
Brief Title: A Comparison of the Effectiveness of Two Approaches in Achieving Smoking Abstinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. LI William Ho Cheung, Principal Investigator, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GOPC
Record Dates: First submitted 2016-02-26; First posted 2016-03-08 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Smoking
Keywords: smoking cessation
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- quit immediately (QI) (Experimental): Subjects in the QI group will receive a smoking cessation booklet plus a brief intervention using the AWARD model: (a) Ask about smoking history, (b) Warn about the high risk, (c) Advise to quit now, as quitting can greatly reduce risks, (d) Refer smokers to a smoking cessation clinic, and (e) Do it again: repeat the intervention during each telephone follow-up. The whole intervention will be limited to less than 1 min or slightly longer if necessary. For the subsequent telephone follow-ups at 1, 3, 6 and 12 months, the counsellor will congratulate to the subjects who successfully quit smoking, while deliver the same brief intervention as a booster for those who continue to smoke.
  Interventions: Behavioral: quit immediately (QI)
- cut down to quit (CDTQ) (Experimental): Subjects in the CDTQ group will also receive the smoking cessation booklet plus a brief intervention using the AWARD model. Instead of asking them to quit immediately, they will be advised gradually cutting down on their cigarette consumption. Also, the subjects will be provided with an education card that contains reduction strategies and a suggested plan to reduce smoking. For the subsequent telephone follow-ups at 1, 3, 6 and 12 months, the nurse counsellor will repeat the warning message that one out of two smokers will be killed by smoking, and remind the subjects of their next reduction target. The counsellor will congratulate subjects who quit or reduce smoking on their success. When subjects fail to quit or reduce their cigarette consumption, the counsellor will reinforce the health hazards of continued smoking and the benefits of quitting, and encourage them to try again immediately or in the near future.
  Interventions: Behavioral: cut down to quit (CDTQ)

INTERVENTIONS:
Behavioral: quit immediately (QI) — advise to quit immediately using the AWARD model
  Arms: quit immediately (QI)
Behavioral: cut down to quit (CDTQ) — advise to reduce cigarette consumption and quit eventally using the AWARD model
  Arms: cut down to quit (CDTQ)

SUMMARY:
The purpose of this study is to test the effectiveness of negotiating self determination to reduce cigarette consumption. A single-blinded multi-centre randomized controlled is employed.

DETAILED DESCRIPTION:
Introduction:

A brief intervention with a small to moderate effect size can potentially benefit a large number of smokers and increase smoking cessation within the community if it is carried out routinely in clinical practices by all or most healthcare professionals or people with minimal training. It is also the most cost-effective smoking cessation programme, because no extra or minimal funding is needed to provide the venue, manpower, and other expenses (but incentives or payments to healthcare professionals and follow-up support would be needed). There is no evidence that longer interventions are more effective than shorter interventions. Brief cessation interventions have been shown to be effective with strong evidence from the investigators' randomised controlled trials and in systematic reviews.

The negotiating self-determination to reduce cigarette consumption is guided by social cognitive and self-determination theories. According to social cognitive theory, self-efficacy is an important personal determinant of human behaviour and has been defined as the belief in one's capability to engage in behaviour to solve difficult tasks. This belief influences decisions on whether a certain form of behaviour will be adopted and maintained. Because self-efficacy is built on a successful experience of overcoming challenging tasks, smokers who have more successful experiences in reducing cigarette consumption tend to have higher levels of self-efficacy. Some evidence has shown that a reduction in smoking may lead to greater self-efficacy to resist smoking, which could increase subsequent quitting. According to self-determination theory, autonomy is another influential determinant of behaviours which is emphasized by freedom of choice. Studies have shown that patients having an opportunity to decide on their own treatment may feel more eager to comply with instructions. The subjects in this study will be allowed to select their own schedules of smoking reduction after the negotiation with the counsellor, such as the percentage of smoking reduction over an acceptable period of time. It is anticipated that the subjects will show more willingness to adhere to their own schedule as a result of an increase in autonomy. Moreover, some evidence has shown that autonomy is positively associated with competence; that is, people have greater autonomy demonstrate higher competence in achieving behavioural change. Consequently, autonomy will facilitate their gradual reduction or cessation of smoking. Most importantly, as a result of reducing the cigarette consumption and lowering down the nicotine dependence, it would be much easier for such smokers to further reduce or quit.

Methods:

Chinese patients attending the general out-patient clinics in Hong Kong for routine follow-up visits who fulfil the following inclusion criteria will be invited to participate in the study.

All smoking patients will be approached by a nurse counselors.

Analysis:

Data analysis will be performed using the Statistical Package for Social Science. In particular, we will use inferential statistics (independent-samples t-test and χ2 test) to examine the homogeneity between the QI and CDTQ groups. We will conduct logistic regression analyses to calculate the odds ratio (OR) and 95% confidence interval (CI) for smoking outcomes, i.e. self-reported and biochemical validated quit rates, self-reported smoking reduction rates and number of quit attempts. We will apply mixed between-within subjects analysis of variance (ANOVA) to determine whether CDTQ is more effective than QI in enhancing self-efficacy (perceived importance, difficulty and confidence) for quitting smoking. We shall adopt the principle of intention to treat. Subjects who are lost to follow-up, refuse to participate in biochemical validations, or withdraw from the study are considered unable to quit or reduce smoking. Depending on the amount and distribution of missing data, other methods, e.g. sensitivity analysis and multiple imputation technique will be used if necessary.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 years or above,
2. smoke at least two cigarettes per day,

Exclusion Criteria:

1. those with unstable medical conditions as advised by the doctor in charge,
2. poor cognitive state or mental illness,
3. participation in other smoking cessation programmes or services.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
self-reported 7-day point prevalence of abstinence | 6 months
self-reported 7-day point prevalence of abstinence | 12 months
self-reported reduction of ≥ 50% in cigarette consumption | 6 months
self-reported reduction of ≥ 50% in cigarette consumption | 12 months

SECONDARY OUTCOMES:
biochemically validated abstinence (exhaled CO test & saliva cotinine test) | 6 months
biochemically validated abstinence (exhaled CO test & saliva cotinine test) | 12 months
self-efficacy in quitting | 6 months
self-efficacy in quitting | 12 months
number of quit attempts made | 6 months
number of quit attempts made | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: William, Ho Cheung Li, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Sai Ying Pun Jockey Club General Out-patient Clinic in Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided